CLINICAL TRIAL: NCT02075970
Title: Optimized EPO Treatment of Neonatal Anemia
Brief Title: Optimized Erythropoietin (EPO) Treatment
Acronym: OETNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John A Widness (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, John A Widness, Professor, Department of Pediatrics, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201306729; 3P01HL046925 (NIH)
Record Dates: First submitted 2013-05-30; First posted 2014-03-03 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Anemia
Keywords: Neonatal; Anemia; Transfusion; Erythropoetin; Epoetin Alpha; Red Blood Cell; Survival; Pharmacodynamics; Model
MeSH Terms: conditions — Anemia, Neonatal; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Epoetin Alpha study 1 (Experimental): Epoetin Alpha Tthe number of separate doses (per kg) to be given over 4 weeks by day of age will not exceed 10. These will be administered as follows: day of life (DOL) 2 (1200 U), DOL 4 (600 U), DOL 5 (600 U), DOL 6 (600U), DOL 7 (600 U), DOL 9 (600 U), DOL 14 (600 U), DOL 15 (600 U), DOL 16 (1200 U), and DOL 28 (600 U). The greatest dose in any 1 wk period is 3600 U.
  Infant study 1 Drug Intervention: all infants will be treated with Epoetin Alpha during the first four weeks of life to provide data for determining: 1) the PK/PD model determined optimized Epoetin Alpha dosing schedule; and 2) clinical and laboratory covariates predictive of which infants are good and poor Epoetin Alpha responder.
  Interventions: Drug: Epoetin Alpha
- Epoetin Alpha study 2 (Placebo Comparator): Epoetin Alpha dosing schedule will be determined based on the results of Infant Study 1.
  Infant Study 2 is a randomized, masked study to test the hypothesis that optimized Epoetin Alpha treatment of VLBW infants predicted to be good responders will result in the elimination of RBCTx relative to poor responders.
  Infant Study 2 in Years 4 and 5 will make use of the knowledge acquired in Infant Study 1 to test the central hypothesis that RBCTX can be eliminated in the majority of good Epoetin Alpha responders by optimal administration of Epoetin Alpha, but only marginal reductions in RBCTx will occur in the poor Epoetin Alpha responders.
  Interventions: Drug: Epoetin Alpha
- Biotinylated red blood cells (Experimental): Individual fetal RBC lifespans will be determined by administering biotinylated red blood cells, both autologous and allogeneic, simultaneously. Left over red blood cells are examined to determine red cell survival.
  Interventions: Drug: Biotinylated Red Blood Cells

INTERVENTIONS:
Drug: Epoetin Alpha — Infant study 1: VLBW infant study subjects (weighing 1.0 to 1.5 kg at birth) who are otherwise receiving standard clinical care will be treated with Epoetin Alpha according to a dosing algorithm.
  Infant study 2:
  Dosing algorithm will be determined by results of Infant Study 1.
  Other Names: Procrit
  Arms: Epoetin Alpha study 1; Epoetin Alpha study 2
Drug: Biotinylated Red Blood Cells — Biotinylated red blood cells will be transfused to infants to determine red blood cell lifespan.
  Other Names: BioRBC
  Arms: Biotinylated red blood cells

SUMMARY:
Neonatal anemia is the most commonly encountered hematologic problem among all neonates cared for in the neonatal intensive care unit (NICU). This project seeks to better understand the pathophysiology and treatment of this challenging and important condition, especially as it affects premature, critically ill very low birth weight (VLBW) infants who require intensive laboratory blood monitoring leading to the need for multiple red blood cell (RBC) transfusions (RBCTX). In the research strategy proposed in Study 1, Aims 1, 2 and 3, recombinant human erythropoietin (Epoetin Alpha, PROCRIT, provided by Janssen Scientific Affairs) will first be administered to 1.0 to 1.5 kg VLBW infants; then comprehensive pharmacokinetics (PK) and pharmacodynamics (PD) data will be systematically gathered and analyzed to identify clinical and laboratory covariate parameters differentiating the infants based on their level of Epoetin Alpha responsiveness. Finally the Epoetin Alpha responsiveness predictors thus determined will be applied prospectively in the Aim 4 Study, a 2 x 2 design in which VLBW infants will be identified as good or poor Epoetin Alpha responders, based on the predictors, and then randomly assigned to receive Epoetin Alpha treatment or no treatment. This will test the central hypothesis: RBCTX can be eliminated in the majority of good Epoetin Alpha responders by optimal administration of Epoetin Alpha, but only marginal reductions in RBCTx will occur in the poor Epoetin Alpha responders. This project challenges the prevailing thinking that the efficacy of Epoetin Alpha dosing in stimulating erythropoiesis is insufficient to eliminate the need for RBC transfusions in VLBW infants. Based on extensive preclinical and clinical PK/PD studies by our PPG team, we contend that previous Erythropoietin treatment studies in VLBW infants were not able to realize the full potential of Erythropoietin to eliminate RBCTX (in contrast to the very successful use of Erythropoietin in adult renal failure patients) because previous VLBW studies were conducted 1) without Epoetin Alpha dosing individualized for the complexities of neonatal erythropoiesis and PK/PD of Epoetin Alpha and 2) without consistent criteria for RBC transfusion, Epoetin Alpha dosing, and patient enrollment. Net Epoetin Alpha responsiveness as reflected in Hb level depends on two components: Epoetin Alpha PD and RBC lifespan (Fig 15). By determining RBC lifespan, we will explain inter-subject variability of Epoetin Alpha responsiveness resulting from one of these components. The fetal lifespan data will be examined for its correlation with gestational age. If the correlation is statistically significant, gestational age will be included in the final selection of covariates for the population PK/PD model to be developed at the end of Infant Study 1. To fully understand the correlation of RBC lifespan with gestational age infants ranging from 22-42 weeks gestational age will be studied. The overall impact of Project 1 will be significant and potentially transformative: the development of a personalized, mechanism-driven approach built on sound principles will improve understanding of neonatal anemia and will be applicable to the care of premature, anemic infants.

RELEVANCE Project 1 results confirming our hypothesis that PK/PD optimized Epo treatment is effective in eliminating RBC transfusions administered to a select sub-group of NICU infants will provide fundamental knowledge about neonatal anemia that will reduce the burden of illness and disability caused by this condition. In addition, our results will stimulate researchers to extend our findings to other sub-groups with neonatal anemia, ie, smaller and sicker infants, and will stimulate novel treatments with similar, new biotechnology-produced protein drugs.

DETAILED DESCRIPTION:
SPECIFIC AIMS Erythropoietin (Epo) stimulates red blood cell (RBC) production. Erythropoietin treatment of anemic, very low birth weight (VLBW) preterm infants has not been as effective as originally anticipated in eliminating multiple RBC transfusions (RBCTX). This conclusion is based on Epoetin Alpha dosing studies employing inconsistent RBCTX criteria, and study designs that did not fully consider Epoetin Alpha's complex pharmacokinetics (PK) and pharmacodynamics (PD). The hypothesis of this project challenges the conclusion that Epoetin Alpha therapy cannot reduce RBCTX in VLBW infants to a clinically important extent. This challenge is based on our novel comprehensive determinations of the PD of endogenous Epo in VLBW infants, and on our recent computer Epo simulation modeling results predicting that RBCTX can be eliminated in a select group of VLBW infants.

Study Objective To develop a pharmacodynamically-based, individualized medicine approach capable of completely eliminating RBCTX in an identifiable group of VLBW infants by optimally administering Epoetin Alpha.

Central Hypotheses Infants with good Epoetin Alpha responsiveness can be identified by a mechanism-driven, individualized prediction model. Optimized Epoetin Alpha treatment of the predicted good responders that is based on sound, evidence based PK/PD principles will eliminate the need for RBCTX.

Epoetin Alpha responsiveness is determined by two key components: 1) RBC production, which depends on Epoetin Alpha PD. 2) RBC lifespan. Individualized covariate-based (ie, patient specific characteristics) prediction of these two components is critical for the development of an individualized prediction model of Epoetin Alpha responsiveness that will be used for testing the Central Hypothesis. These important predictors of Epoetin Alpha responsiveness will be investigated in the following Specific Aims (SA) and Hypotheses (HY):

INFANT STUDY 1 (Years 1-3) performed in VLBW infants with birth weights from 1.0 to 1.5 kg SA 1 Determine clinical and laboratory covariates (ie, patient-specific characteristics) controlling the large inter-subject variability in Epoetin Alpha's PD using data from Epoetin Alpha dosing of VLBW infants HY 1 The inter-subject variability in Epoetin Alpha's PD is predictable by several covariates that are identifiable by our PK/PD modeling approach.

SA 2 Determine the lifespan of fetal RBC in the gestational age spectrum of the study infants.

HY 2 There exists a significant inter-subject variability in the lifespan of fetal RBCs in VLBW infants that is predictable based on gestational age.

SA 3 Derive an individualized, optimal Epoetin Alpha dosing algorithm and an individualized prediction model for the Epoetin Alpha responsiveness in VLBW infants from the results in Specific Aims 1 and 2.

HY 3 Crossvalidation-type computer simulations based on individualized and optimized Epoetin Alpha dosing in a subgroup of VLBW infants with good Epoetin Alpha responsiveness, identified by the prediction model, will indicate that RBCTX can be avoided in a select group of VLBW infants.

INFANT STUDY 2 (Years 3-4, to be addressed as a modification after completion of study 1) also performed in VLBW infant with birth weights from 1.0 to 1.5 kg SA 4 Apply the optimal Epoetin Alpha dosing algorithm and Epoetin Alpha responsiveness prediction model developed in Infant Study 1 to an Epoetin Alpha dosing study to test the Central Hypothesis.

HY 4 The subgroup of VLBW infants with good Epoetin Alpha responsiveness will have a higher proportion of infants that will not have any RBCTX compared to those with poor Epoetin Alpha responsiveness.

Expected Outcomes SA 1 Among the covariates considered in Specific Aims 1 (e.g. clinical neonatal/maternal factors, blood cell parameters, cytokines linked to erythropoiesis, inflammation biomarkers, oxidative stress, iron status, and genetic factors), we will identify several with statistically significant correlations to Epoetin Alpha's PD.

SA2 The lifespan of fetal RBCs will show similar relationship to gestational age as that which was observed by us in the ovine fetus.

SA3 The model will accurately predict individual Epoetin Alpha responsiveness to optimized Epo dosing and will provide strong support for our hypothesis that RBCTX can be completely eliminated in a select group of VLBW infants.

SA4 Infant Study 2 will show that the select group of VLBW infants that are predicted to be good Epoetin Alpha responders by the combined use of an individualized Epoetin Alpha responsiveness prediction model and an optimal, individualized Epo dosing algorithm will have a greater proportion of infants who do not require any RBCTX compared to those predicted to have poor Epoetin Alpha responsiveness.

A successful completion of the proposed research is potentially transformative and is likely to be applied to the care of VLBW infants, resulting in a significant overall impact. Moreover, a successful demonstration of the utility and power of these principles will lead to improvements in the complex pharmacotherapy of VLBW infants, who are among the most difficult to study of any patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menstrual age at birth less than 37 wk;
2. birth weight of 1,001 to 1,500 g;
3. postnatal age <48 h;
4. respiratory distress requiring ventilation;
5. signed consent by parent or guardian.

Exclusion Criteria:

1. Anticipated survival <72 h;
2. Hemolytic anemia due to alloimmune disease (including due to ABO), and other hemolytic disease processes;
3. Major anomalies that are life-threatening during the neonatal and infant periods (central nervous system, cardiac, metabolic chromosomal including, but not limited to, trisomies, deletions, and trinucleotide repeats);
4. Clinical seizures;
5. Congenital thrombotic or hemorrhagic conditions including disseminated intravascular coagulation;
6. Positive blood or spinal fluid bacterial or fungal culture, or other laboratory and/or clinical data indicative of sepsis, including TORCH infections, prior to 48 h of age;
7. Hematocrit >50%;
8. Platelet count >400,000 per µL in first 48 h of life;
9. Hypertension with systolic blood pressure >100 mm Hg.
10. Any condition, in the opinion of the investigators, that would compromise the well being of the subject or the study, or prevent the subject from meeting or performing study requirements.

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of red blood cell transfusions | From date of randomization through day of life 28 or death, whichever comes first
  The count of the number of packed red blood cell transfusions an infant receives during the entire course of their initial hospital stay.

SECONDARY OUTCOMES:
Survival of Fetal Red Blood Cells in number of days | From date of transfusion of biotinylated red blood cells until biotinylated red blood cells are no longer detectable in leftover blood samples, or death, whichever comes first. An expected average of 80-120 days. Assessed up to 5 months.
  The count of the number of days that biotinylated red blood cells are identified in leftover blood samples. Counted from the day of transfusion until they are no longer able to be identified.

OTHER OUTCOMES:
Derivation of an individualized, optimal Epoetin Alpha dosing algorithm and prediction model for each subject | From birth through discharge or death, whichever comes first. An average of 4 weeks to 6 months. Assessed up to 12 months.
  Using the covariates, red cell transfusions, blood loss due to labs, and growth, a model will be developed that will accurately predict individual Epoetin Alpha responsiveness to optimized Epoetin Alpha dosing.

CONTACTS AND LOCATIONS:
Overall Officials: John A Widness, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No